CLINICAL TRIAL: NCT02892838
Title: Should my New Knee Rotate? A Randomised, Controlled Clinical Trial to Compare Fixed and Mobile Bearing Total Knee Arthroplasties Using the SCORPIO PS and SCORPIO+ PS Knee Systems
Brief Title: Should my New Knee Rotate?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC02-055
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2016-07

CONDITIONS: Arthritis of the Knee Joint
Keywords: mobile bearing knee prosthesis
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mobile bearing knee prosthesis (Experimental): use of the Scorpio mobile bearing knee system for total knee arthroplasty
  Interventions: Device: mobile bearing knee system for total knee arthroplasty
- fixed bearing (Active Comparator): use of the Scorpio fixed bearing knee system for total knee arthoplasty
  Interventions: Device: fixed bearing total knee prosthesis

INTERVENTIONS:
Device: mobile bearing knee system for total knee arthroplasty
  Arms: mobile bearing knee prosthesis
Device: fixed bearing total knee prosthesis
  Arms: fixed bearing

SUMMARY:
Total Knee Arthroplasty (TKA) is the surgical reconstruction of the knee joint in order to relieve pain, restore function and correct deformity. It is a very common surgical procedure with figures showing more than 500'000 arthroplasties performed annually worldwide. Total knee arthroplasty is considered one of the most successful types of joint reconstruction in that surgical results usually meet and even exceed expectations. Much of the current literature focuses on the issues relating to implant wear as a potential failure mode for artificial knee implants. It has been suggested that knee with mobile or rotating bearing options, such as the comparative device proposed for this clinical investigation, may survive longer than fixed bearing knee designs because of the greater contact surface area possible with more congruent components with unconstrained, mobile component design.

DETAILED DESCRIPTION:
This is a prospective, comparative, randomised, open-label, single center, multiple surgeons clinical study. The Scorpio PS Superflex and the Scorpio PS mobile bearing are to be implanted for evaluation in this study. Patients will be randomised to one of two equal sized groups. In the first group patients will be treated with the Scorpio PS Superflex, whilst in the second group patients will be treated with the Scorpio PS mobile bearing implant.

Evaluations consist of the KSS score, Chair rise and stair climb tests, radiology assessments, patient questionnaires, at multiple timepoints: pre-operative, 6 weeks, 3 months, 6 months 1 year, 2 years and 5 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring cemented primary total knee replacement.
* Patients with a diagnosis of osteoarthritis (OA), avascular necrosis (AVN) or post-traumatic arthritis (TA)
* Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographic evaluations and the prescribed rehabilitation.
* Patient who have intact collateral ligaments.
* Patient who signed the Ethics Committee approved specific Informed Consent Form prior to surgery.

Exclusion Criteria:

* Patient where patella will not be resurfaced.
* Patients with active or suspected infection.
* Patients with a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the study (i.e. severe osteoporosis, Paget's disease, renal osteodystrophy) or is immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
* The patient has a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weightbearing or places an extreme load on the implant during the healing period.
* Patients, who as judged by the surgeon, are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2003-09; Primary Completion 2008-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Anterior knee pain during stair rise | 5 years
  Anterior knee pain using VAS during stair rise at different follow up moments until 5 years after surgery
Anterior knee pain during stair climb | 5 years
  Anterior knee pain using VAS during stair climb at different FU moments

SECONDARY OUTCOMES:
passive and active Range of motion | 5 years
  measuring passive and active range of motion (flexion / extension) using a goniometer at different FU moments
patella compression pain | 5 years
  patella compression pain at physical examination at different FU moments defined as yes of no when putting mild pressure on the patella
patient satisfaction | 5 years
  measuring patient satisfaction using the RAND-36 questionnaire at different FU moments

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feczko, MD, Principal Investigator — orthopedic surgeon MUMC Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feczko PZ, Jutten LM, van Steyn MJ, Deckers P, Emans PJ, Arts JJ. Comparison of fixed and mobile-bearing total knee arthroplasty in terms of patellofemoral pain and function: a prospective, randomised, controlled trial. BMC Musculoskelet Disord. 2017 Jun 29;18(1):279. doi: 10.1186/s12891-017-1635-9. PMID 28662692